CLINICAL TRIAL: NCT06920888
Title: Is Less More? Dosing and Sequencing Effects of Cognitive Therapies for Anxiety and Depression
Brief Title: Is Less More? Dosing and Sequencing Effect
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4282-00031B
Record Dates: First submitted 2025-03-17; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Depression/Anxiety
Keywords: CBT; Combinatory effects; MOST; Optimizing; Dosing; Sequencing effects
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Cognitive Restructuring

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of four groups, receiving one or both components (CR [A] and AA [B]) under investigation, all over the course of six sessions of treatment. One group will receive component A for 6 sessions, another group will receive component B for 6 sessions, a third group will receive component A for 3 sessions followed by component B for 3 sessions, and a fourth group will receive component B for 3 sessions followed by component A for 3 sessions. All groups will begin with a 3-week waiting period, thus employing a multiple baseline design.
Who Masked: Participant
Masking Description: Participants will be unaware both of the planned component comparisons and of the study hypotheses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cognitive restructuring (CR) (Experimental): 6 sessions of CR drawn from classic Cognitive Behavioral Therapy (CBT)
  Interventions: Behavioral: Cognitive restructuring
- Attention allocation (AA) (Experimental): 6 sessions of AA building on contemporary CBTs
  Interventions: Behavioral: Attention allocation
- CR followed by AA (Experimental): 3 sessions of CR followed by 3 sessions of AA
  Interventions: Behavioral: Cognitive restructuring; Behavioral: Attention allocation
- AA followed by CR (Experimental): 3 sessions of AA followed by 3 sessions of CR
  Interventions: Behavioral: Cognitive restructuring; Behavioral: Attention allocation

INTERVENTIONS:
Behavioral: Cognitive restructuring — CR drawn from classic CBT
  Arms: AA followed by CR; CR followed by AA; Cognitive restructuring (CR)
Behavioral: Attention allocation — AA drawn from contemporary CBTs
  Arms: AA followed by CR; Attention allocation (AA); CR followed by AA

SUMMARY:
The investigators want to evaluate core components from cognitive behavioral psychotherapies (CBTs) with the aim of investigating dosing and combinatory effects on conditions of anxiety and depression.

DETAILED DESCRIPTION:
In the present study, participants will be randomly assigned to one of four groups, receiving one or both treatment components under investigation, all over the course of six sessions of treatment.

1. It is hypothesized that both component A (Cognitive Restructuring) and component B (External Attention Allocation) will be efficient in reducing symptoms of depression and anxiety when delivered separately, both when delivered over 3 and 6 sessions. The difference between components as well as between the number of sessions on primary and secondary outcomes will be explored.
2. The combinatory effects, comparing the effect of receiving Component A subsequent to Component B and vice versa will be explored.
3. The process of change in both components will be explored.
4. Group differences in participants' experience of being the recipient of the components (either individually or combination) both qualitatively (free descriptions of their experience with using them) and quantitatively (questionnaires concerning the understanding and employment) will be explored.
5. The moderating effect of baseline characteristics including baseline symptomatology, diagnoses, personality functioning, and working alliance will be explored.
6. Potential harmful effects will be explored in each group.

ELIGIBILITY:
Inclusion Criteria:

(i) age ≥ 18 years, (ii) Clinically relevant symptoms of an anxiety disorder (with the exception of specific phobia) and/or depressive disorder according to GAD-7≥10, SIAS ≥37, PHQ-9 ≥10, or PDSS ≥9, (iii) Danish language proficiency, (iv) ability and willingness to give informed consent, (v) no or stable antidepressant/antianxiety medication (i.e., same dosage for ≥ 6 weeks), (vi) access to either a smartphone, tablet, or computer with video camera.

Exclusion Criteria:

(i) severe depression deemed to require more intense psychotherapy or medication (PHQ-9-score of 20 or more combined with a clinical evaluation), (ii) currently receiving other psychotherapy or counseling, (iii) a history of bipolar disorder, (iv) current or past psychotic episode, (v) substance abuse or dependence judged to require treatment, (vi) suicide risk requiring immediate hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | Change from pre (just prior to session 1) to post treatment (after session 6), app. 7 weeks in total.
  Patient Health Questionnaire-9 (Kroenke et al., 2001; Spitzer et al., 1999; Spitzer et al., 2000; PHQ-9). 9 items are rated on a scale from 0 to 3, with a potential total range from 0 to 27. Larger scores mean more depressive symptoms (i.e., a negative outcome).
Anxiety symptoms | Change from pre (just prior to session 1) to post treatment (after session 6), app. 7 weeks in total.
  Beck's Anxiety Inventory (Beck et al., 1988; Beck & Steer, 1991; BAI). 21 items are rated on a scale from 0 to 3 with a total score thus ranging from 0 to 63. A higher score is indicative of more anxiety symptoms (i.e., a negative outcome).

SECONDARY OUTCOMES:
Depressive symptoms | Change from pre treatment (just prior to session 1) through follow-up (6 months after treatment has ended), app. 33 weeks in total.
  PHQ-9
Anxiety symptoms | Change from pre treatment (just prior to session 1) through follow-up (6 months after treatment has ended), app. 33 weeks in total.
  BAI
Symptoms of generalized anxiety disorder | Changes from pre (just prior to session 1) to post treatment (just after session 6) and through follow-up (6 months after treatment has ended) only for those individuals that scores above cut-off during the screening process, app. 33 weeks in total.
  General Anxiety Disorder-7 (Spitzer et al., 2006; GAD-7). 7 items are rated on scale from 0 to 7 with total scores ranging from 0 to 21. Higher scores are indicative of more symptoms of GAD (i.e., a negative outcome).
Symptoms of panic disorder | Changes from pre (just prior to session 1) to post treatment (just after session 6) and through follow-up (6 months after treatment has ended) only for those individuals that scores above cut-off during the screening process, app. 33 weeks in total.
  The Panic Disorder Severity Scale - Self-Report Version (Houck et al., 2002; PDSS-SR). 7 items are rated on a scale form 0 to 4, with total scores ranging from 0 to 28. Higher scores are indicative of more symptoms of panic disorder (i.e., a negative outcome).
Symptoms of social anxiety disorder | Changes from pre (just prior to session 1) to post treatment (just after session 6) and through follow-up (6 months after treatment has ended) only for those individuals that scores above cut-off during the screening process, app. 33 weeks in total.
  The Social Interaction Anxiety Scale (Mattick & Clarke, 1998, SIAS). 20 items are rated on a scale from 0 to 4 with total scores ranging form 0 to 80. Higher scores are indicative of more symptoms of social anxiety disorder (i.e., a negative outcome).
Worry | Changes from pre (just prior to session 1) to post treatment (just after session 6) and through follow-up (6 months after treatment ended), app. 33 weeks in total.
  The Penn State Worry Questionnaire (Meyer et al., 1990; PSWQ). 16 items are rated on a 5-point scale, with total scores ranging from 16 to 75. Higher scores indicate more worry (i.e., a negative outcome).
Decentering | Changes from pre (just prior to session 1) to post treatment (just after session 6) and through follow-up (6 months after treatment ended), app. 33 weeks in total.
  The Experiences Questionnaire (Fresco et al., 2007; EQ), decentering subscale. 11 items are rated on a scale from 1 to 5, with total scores ranging from 11 to 55. Higher scores mean better ability to decenter (i.e., a positive outcome).
Cognitive change | Changes from pre (just prior to session 1) to post treatment (just after session 6) and through follow-up (6 months after treatment ended), app. 33 weeks in total.
  The Cognitive Change - sustained scale (Schmidt et al., 2019; CC). 9 items rated on a scale from 0 to 6 with total scores ranging from 0 to 63. Higher scores mean better ability to employ cognitive change (i.e., a positive outcome).
Cognitive reappraisal | Changes from pre (just prior to session 1) to post treatment (just after session 6) and through follow-up (6 months after treatment ended), app. 33 weeks in total.
  ERQ-reappraisal = Emotion Regulation Questionnaire - reappraisal subscale (Gross & John, 2003; ERQ-r). 6 items are rated on a scale from 1 to 7 with total scores ranging from 6 to 42. Higher scores mean better ability to employ cognitive reappraisal (i.e., a positive outcome).
Mindfulness | Changes from pre (just prior to session 1) to post treatment (just after session 6) and through follow-up (6 months after treatment ended), app. 33 weeks in total.
  Five Facet Mindfulness Questionnaire-15 (Baer et al., 2006; FFMQ-15). 15 items are rated on a scale from 1 to 5 with total scores ranging from 15 to 75. Higher scores mean higher levels of mindfulness (i.e., a positive outcome).
Attention control | Changes from pre (just prior to session 1) to post treatment (just after session 6) and through follow-up (6 months after treatment ended), app. 33 weeks in total.
  The Attention Control Scale (Derryberry & Reed, 2002; ATQ-short form. 10 items are rated on a scale from 1 to 4 with total scores ranging from 10 to 40. Higher scores are indicative of better attention control (i.e., a positive outcome).
Valued Living | Changes from pre (just prior to session 1) to post treatment (just after session 6) and through follow-up (6 months after treatment ended), app. 33 weeks in total.
  Valuing Questionnaire (Smout et al., 2014; VQ). 10 items are rated on a scale from 0 to 6 with total scores ranging from 0 to 60. Higher scores a indicative of actions/life being guided by personally held values (i.e., a positive outcome).
Quality of life (well-being) | Changes from pre (just prior to session 1) to post treatment (just after session 6) and through follow-up (6 months after treatment ended), app. 33 weeks in total.
  the World Health Organization-5 questionnaire (Bech, 1999; Topp et al., 2015; WHO-5). 5 items are rated on a scale from 0 to 5 with total scores ranging from 0 to 25. Higher scores are indicative of higher levels of life quality (i.e., a positive outcome).
Personality functioning | Changes from pre (just prior to session 1) to post treatment (just after session 6) and through follow-up (6 months after treatment ended), app. 33 weeks in total.
  Level of Personality Function Scale-Brief Form 2.0 (Weekers et al., 2019; LPFS-BF). 12 items are rated from 1 to 4 with total scores ranging from 12 to 48. Higher scores are indicative of better personality functioning (i.e., a positive outcome).
Harm/negative effects | Measured only one time, that is, post treatment (just after the 6 sessions).
  The Negative Effects Questionnaire (Rozental et al., 2019; NEQ). 32 questions are answered yes/no. If yes, items are rated on a scale from 1 to 5 and participants are asked if the negative effect experience can be attrubuted to the treatment or other crcumstances. Total scores range from 32 to 160 with higher scores indicating more negative effects (i.e., a negative outcome).
Information overload | Measured only one time, that is, post treatment (just after the 6 sessions).
  Information Overload scale (adapted from Jensen et al., 2014; IO). 8 items are rated from 1 to 4 with total scores ranging from 8 to 32. Higher scores are indicative of more information overload (i.e., a negative outcome).

OTHER OUTCOMES:
Depressive symptoms | Session-by-session changes from pre-treatment (just prior to session 1) to post-treatment (just after 6 sessions), app. 7 weeks in total.
  PHQ-9, rated as noted above.
Anxiety symptoms | Session-by-session changes from pre-treatment (just prior to session 1) to post-treatment (just after 6 sessions), app. 7 weeks in total.
  BAI, rated as noted above.
Decentering | Session-by-session changes from pre-treatment (just prior to session 1) to post-treatment (just after 6 sessions), app. 7 weeks in total.
  EQ, rated as noted above.
Cognitive change | Session-by-session changes from pre-treatment (just prior to session 1) to post-treatment (just after 6 sessions), app. 7 weeks in total.
  CC (5 items), rated as noted above but only five items are evaluated on a session-by-session basis.
Cognitive reappraisal | Session-by-session changes from pre-treatment (just prior to session 1) to post-treatment (just after 6 sessions), app. 7 weeks in total.
  ERQ-r, rated as noted above.
Mindfulness | Session-by-session changes from pre-treatment (just prior to session 1) to post-treatment (just after 6 sessions), app. 7 weeks in total.
  FFMQ-15, rated as noted above.
Attention control | Session-by-session changes from pre-treatment (just prior to session 1) to post-treatment (just after 6 sessions), app. 7 weeks in total.
  ATQ-short, rated as noted above.
Strategy use | Session 3 [app. week 3 of the intervention] and session 6 [app. week 6 of the intervention] (the measure is only obtained at those two time points).
  Description [free text] of a situation in the past week where participants used or could have used the treatment component (CR or AA). Individuals in the combined arms (receiving both components) will also describe [free text] how they see themselves using the two strategies.
Experience of therapy | Session-by-session changes from pre-treatment (just prior to session 1) to post-treatment (just after 6 sessions), app. 7 weeks in total.
  The participant will report on 1) the extent to which the individual understands the treatment component, 2) how competent they feel about being able to apply the treatment component in everyday life, 3) how useful they consider the treatment component to be, 4) how much they want to use the component, and 5) how often they actually used the treatment component in everyday life.
  They will do so retro and prospectively and for both components when relevant.
Working alliance | Measure obtained two times; at session 2 [app. week 2 of the intervention] and session 4 [app. week 4 of the intervention].
  Working Alliance Inventory - Short Revised (Munder et al., 2010; WAI-SR). 12 items rated on a scale from 1 to 5 with total scores ranging from 12 to 60. Higher scores indicate better working alliance (i.e., a positive outcome).